CLINICAL TRIAL: NCT06063993
Title: Evaluation of Pulse-oximetry Derived Perfusion Index Change Post Passive Leg Raising for Fluid Responsiveness in Critically Ill Patients
Brief Title: Evaluation of Perfusion Index Change Post Passive Leg Raising for Fluid Responsiveness in Critically Ill
Status: Completed | Type: Observational
Sponsor: National Hepatology & Tropical Medicine Research Institute (Other Government)
Responsible Party: Principal Investigator, ICU, fellow of intensive care medicine, National Hepatology & Tropical Medicine Research Institute
Other Study IDs: 27-2023
Record Dates: First submitted 2023-08-28; First posted 2023-10-03 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Fluid Responsiveness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Peripheral Perfusion Index (PI) has been investigated for its use in hemodynamic monitoring. The PI is derived from the photoelectric plethysmographic signal of the pulse oximeter. The changes in the PI reflect changes in peripheral vasomotor tone.

In critically ill patients, the same value was found to represent a very sensitive cutoff point for determining abnormal peripheral perfusion, as defined by a prolonged Capillary Refill Time (CRT). However, age, gender, and ambient temperature have all been shown to affect the measure of CRT in normal volunteers, and the presence of a CRT > 2 or 3 seconds was not predictive of blood loss in phlebotomized volunteers. In addition, the CRT has been shown to have poor intra-observer agreement when a cutoff a two seconds was used in adult emergency room patients.13 Therefore, PI can be used for monitoring peripheral perfusion in critically ill patients.14PI shows the perfusion status of the tissue in the applied area for an instant and a certain time interval. The PI value ranges from 0.02% (very weak) to 20% (strong).

As non-invasive CO monitors (ICON ®) is not available in many centers in our country due to its high cost, we try to validate other simple non-invasive method to be used to assess FR in critically ill patients.

The purpose of this study is to investigate the efficacy of pulse-oximeter derived PI measurement in assessment of fluid responsiveness in critically ill patients in comparison with CO response.

DETAILED DESCRIPTION:
After approval by NHTMRI-IRB Ethical Committee.All demographic data will be obtained including the patients age, sex,associated co-morbidities (diabetes mellitus & hypertension).

Continuous blood pressure, continuous electrocardiogram, heart rate (HR), and SpO2 (measured by pulse oximetry).

Patients who are eligible and have signs of hemodynamic instability, PLR will be performed by adjusting the bed and not by manually raising the patient's legs. Bronchial secretions must be carefully aspirated before PLR. If awake, the patient should be informed of what the test involves.PLR should start from the semi-recumbent and not the supine position. Adding trunk lowering tosupine position and leg raisingfor 45° for 60 seconds, this mobilizes venous blood from the large splanchnic compartment, thus magnifying the increasing effects of leg elevation on cardiac preload.18COand PI measurements will be recorded in the same patients.

ELIGIBILITY:
Inclusion Criteria:

* The subjects are adults aged ≥18 years old
* admitted tothe intensive care unit of the National Hepatologyand Tropical Medicine Research Institute (NHTMRI).
* Patients with clinical signs of hemodynamic instability i.e. a systolic blood pressure < 90 mmHg or decrease in systolic blood pressure > 40 mmHg, signs of organ hypoperfusion as oliguria < 0.5ml/Kg/hour.

Exclusion Criteria:

* If there is known peripheral vascular disease
* or ≥ 2 vasopressors with the maximum doses
* or in the presence of nail polish as readings from pulse oximeter will be distortedin these cases
* or if there is contraindication for PLR as uncontrolled hemodynamic status
* intracranial hypertension
* severe chronic obstructive pulmonary disease
* broncho-alveolar fistula
* severe emphysema
* and those with pre-existing comorbidities including severe left and right ventricular dysfunction, severe pulmonary hypertension
* severe obesity (BMI >40 kg/m2)
* pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be subdivided into two groups; responders and non-responder:
  * Responders group 1 (R); were defined as those who had increase of 10% in CO from baseline measured by EC after PLR.
  * Non-responders group 2 (NR); those who had increase of less than 10% in CO from baseline measured by EC after PLR.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
Fluid responsiveness | during PLR passive leg raising during 60 seconds
  to detect reliability of PI to detect Fluid responsiveness (FR) in critically ill patients

SECONDARY OUTCOMES:
PI reliability | by the end of statistical analysis of the study up to one year
  obtain the sensitivity and specificity of this index for FR.

CONTACTS AND LOCATIONS:
Locations (1):
- NHTMRI, Cairo, Egypt